CLINICAL TRIAL: NCT01290198
Title: Role of Epoxy-eicosatrienoic Acids in Post-occlusive Hyperemia and Thermal Hyperemia
Acronym: EETY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: DCIC 10 01
Record Dates: First submitted 2011-02-03; First posted 2011-02-04 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Healthy Volunteers
Keywords: epoxy-eicosatrienoic acid; Laser Doppler; Endothelium derived hyperpolarizing factor; cutaneous microcirculation; post-occlusive hyperaemia; thermal hyperemia; intradermal microdialysis; fluconazole
MeSH Terms: interventions — NG-Nitroarginine Methyl Ester; omega-N-Methylarginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vehicle without ANESDERM (lidocaine, prilocaine) (Placebo Comparator)
  Interventions: Drug: Microdialysis of fluconazole, vehicle and N(G)-nitro-L-arginine-methyl ester (L-NMMA)
- Vehicle with ANESDERM (lidocaine, prilocaine) (Active Comparator)
  Interventions: Drug: Microdialysis of fluconazole, vehicle and N(G)-nitro-L-arginine-methyl ester (L-NMMA)
- Fluconazole without ANESDERM (lidocaine, prilocaine) (Active Comparator)
  Interventions: Drug: Microdialysis of fluconazole, vehicle and N(G)-nitro-L-arginine-methyl ester (L-NMMA)
- Fluconazole with ANESDERM (lidocaine, prilocaine) (Active Comparator)
  Interventions: Drug: Microdialysis of fluconazole, vehicle and N(G)-nitro-L-arginine-methyl ester (L-NMMA)

INTERVENTIONS:
Drug: Microdialysis of fluconazole, vehicle and N(G)-nitro-L-arginine-methyl ester (L-NMMA) — At the first three visits, volunteers will receive fluconazole (650µmol/L and 6.5mmol/L) and vehicle (NaCl 0.9%), and at the fourth, these plus L-NMMA (10mmol/L), delivered by microdialysis in the forearm, with or without anesthesia. Then post-occlusive hyperemia and thermal hyperemia are performed.

SUMMARY:
The objective of this proof of concept study is to assess the involvement of epoxy-eicosatrienoic acids (EETs) in post-occlusive hyperemic and thermal hyperemia responses, and the interaction between nitric oxide (NO) and EETs, using the latest methods for the study of functional microcirculation.

DETAILED DESCRIPTION:
The EETY study is a single-center proof of concept study in healthy volunteers. The main objective is to study the involvement of epoxy-eicosatrienoic acids (EETs) in the reactivity of cutaneous microcirculation during post-occlusive hyperemia and thermal hyperemia, by studying the response to microdialysis of fluconazole (an inhibitor of EETs) versus control, on the forearm.

Response is measured by the amplitude of the post-occlusive hyperemia and thermal hyperemia peaks (maximum amplitude as a percentage of maximal vasodilation and areas under the curve: AUC) during the injection of fluconazole compared to an intradermal injection of solvent (NaCl 9 ‰).

The subjects are healthy volunteers of both sexes, aged between 18 and 35, non-smokers and in good health. Over two years, 30 subjects will be included in the study for 6 to 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35 years
* Affiliated to the French social security system or beneficiary a similar regime
* In good health

Exclusion Criteria:

* Active smoker
* Pregnant, parturient, breast-feeding
* Person deprived of civil liberties by judicial or administrative measure; person under legal protection,
* Minor less than 18 years
* Within period exclusion for other clinical research studies
* Person has exceeded the annual compensation for participation in trials
* Person with active disease or with prolonged treatment, excluding oral contraceptives and paracetamol
* Asthma, urticaria, angioedema, known drug allergy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-02; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Amplitude of the post-occlusive hyperemia and thermal hyperemia following the injection by intradermal microdialysis of fluconazole compared with injection of vehicle (NaCl 9 ‰) | 2 hours
  maximum amplitude as a percentage of maximal vasodilation and area under the curve: AUC

SECONDARY OUTCOMES:
Amplitude of the post-occlusive hyperemia and thermal hyperemia following the injection by intradermal microdialysis of fluconazole, at 2 concentrations, or vehicle (NaCl 9 ‰) | 2 hours
  maximum amplitude expressed as percentage of maximal vasodilation and AUC
Amplitude of the post-occlusive hyperemia and thermal hyperemia following the injection by intradermal microdialysis of fluconazole or vehicle (NaCl 9 ‰), with and without ANESDERM ® (lidocaine, prilocaine) | 2 hours
  maximum amplitude expressed as percentage of maximal vasodilation and AUC
Amplitude of the post-occlusive hyperemia and thermal hyperemia following the injection by intradermal microdialysis of fluconazole or vehicle (NaCl 9 ‰), with and without N(G)-nitro-L-arginine-methyl ester (L-NMMA) | 2 hours
  maximum amplitude expressed as percentage of maximal vasodilation and AUC

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Cracowski, MD,PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Clinical Pharmacology Unit, Grenoble, France